CLINICAL TRIAL: NCT06008925
Title: A Dose Ascending, Open Phase Ib/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of VG161 Combined With Nivolumab Injection in Subjects With Metastatic Gastric Cancer
Brief Title: Clinical Study of VG161 Combined With Nivolumab Injection in Patients With Advanced Metastatic Gastric Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CNBG-Virogin Biotech (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG161-C202
Record Dates: First submitted 2023-03-05; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Gastric Cancer
Keywords: Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Part1:
  VG161:
  1) 1.0 × 10 ^ 8 PFU daily on Day 1 of each cycle (D1); 2)1.0 × 10 ^ 8 PFU daily for 2 consecutive days on Days 1-2 of each cycle (D1-D2); 3)1.0 × 10 ^ 8 PFU daily for 3 consecutive days on days 1-3 (D1-D3) in the first cycle; 1.0 × 10 ^ 8 PFU daily for 2 consecutive days on days 1-2 (D1-D2) in the second and subsequent cycles; Nivolumab Injection: 3 mg/kg every 2 weeks (D8, D22)
  Part2:
  Depends on the recommended dose in Part1
  Interventions: Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)); Drug: Nivolumab Injection

INTERVENTIONS:
Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)) — Intratumoral injection only. Dosing days may be Day 1 or Days 1-3 only.
  Other Names: VG161
Drug: Nivolumab Injection — Administered once at 3 mg/kg intravenously on Days 8 and 22 of each cycle.
  Other Names: OPDIVO

SUMMARY:
VG161 is a recombinant human-IL12/15/PDL1B oncolytic HSV-1 injection. This study will be conducted in combination with nivolumab injection in HSV seropositive subjects with advanced metastatic gastric or gastroesophageal junction adenocarcinoma who have previously received two or more systemic treatment regimens (which must include anti-PD-1 monoclonal antibodies). This is an open-label study divided into two parts.

Part 1: This part is an escalating dose trial to explore the safety of the combination and determine the recommended safe dose of the combination.

Part 2: This part is an extension trial to investigate the preliminary efficacy of the combination at a safe dose.

DETAILED DESCRIPTION:
Part1(Phase Ib primary objective): To evaluate the safety and tolerability of VG161 administered by intratumoral injection combined with Nivolumab Injection in the treatment of patients with advanced metastatic gastric or gastroesophageal junction adenocarcinoma who have previously received two or more systemic treatment regimens (including anti-PD-1 monoclonal antibodies), explore the most suitable recommended Phase II dose (RP2D) for combination therapy, and determine the recommended regimen for combination therapy in Phase IIa clinical trials. Secondary objectives: 1) To preliminarily evaluate the antitumor activity of VG161 combined with nivolumab injection in the treatment of patients with advanced gastric cancer; 2) To monitor the changes of immunological parameters related to pharmacodynamics; 3) To evaluate the relevant immunological characteristics of tumor biopsy samples; 4) To evaluate the pharmacokinetic (PK) characteristics and viral excretion of single and multiple intratumoral injections of VG161;

Part2(Phase IIa Primary Objective): To further evaluate the safety and efficacy of intratumoral injection of VG161 combined with nivolumab injection in patients with advanced metastatic gastric or gastroesophageal junction adenocarcinoma who have previously received two or more systemic treatment regimens (which must include anti-PD-1 monoclonal antibodies), with the primary outcome measure of efficacy being objective response rate (ORR). Secondary objectives: 1) To evaluate the secondary outcome measures of the efficacy of combined treatment; 2) To monitor the pharmacodynamic-related changes in immunological parameters; 3) To evaluate the relevant immunological characteristics of tumor biopsy samples;

ELIGIBILITY:
Inclusion Criteria:

- (Subjects must meet all of the following inclusion criteria to enter the trial)

1. Subjects must give informed consent to this study before the trial and voluntarily sign a written informed consent form.
2. aged 18 to 75 years (inclusive), male or female.
3. Patients with advanced metastatic gastric or gastroesophageal junction adenocarcinoma confirmed by histopathology or cytology.
4. According to the Guidelines for the Diagnosis and Treatment of Gastric Cancer (CSCO, version 2021), patients must have previously failed two or more systemic treatment regimens (which must include anti-PD-1 monoclonal antibodies), or patients who cannot continue treatment due to severe adverse reactions as judged by the investigator.
5. Be able to provide paraffin blocks and/or tissue sections of previously archived pathological tissues, or willing to undergo tumor tissue biopsy before administration.
6. The presence of at least one measurable CT scan according to RECIST 1.1 and meeting the requirements for an acceptable injection dose volume (or the first injection dose volume in Phase IIa) in the current dose group, tumor metastases that can be injected under ultrasound guidance (injected lesions are best major tumor burden lesions), and the baseline longest diameter of the injected lesion (lymph node lesions are short diameters) > 1.5 cm.
7. Positive test result for herpes simplex virus I antibodies (HSV-1 IgG or HSV-1 IgM).
8. ECOG performance status score 0-1.
9. Expected survival time of more than 3 months.
10. adequate organ function: 1) blood routine (no blood transfusion or colony-stimulating factor treatment within 14 days): ANC ≥ 1.5 × 10^9/L, PLT ≥ 100 × 10^9/L, Hb ≥ 85 g/L, lymphocyte count ≥ 1.5 × 10^9/L (for lymphocyte count 0.8 × 10^9/L to 1.5 × 10^9/L, the investigator judged whether to enroll); 2) liver function: TBIL ≤ 1.5 × ULN, ALT ≤ 3 × ULN, AST ≤ 3 × ULN; 3) renal function: Cr ≤ 1.5 × ULN, and creatinine clearance ≥ 45ml/min (calculated according to Cockcroft-Gault formula); 4) coagulation function: activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, international normalized ratio (INR) ≤ 1.5 × ULN.
11. eligible subjects of childbearing potential (men and women) must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) during the trial and for at least 90 days after the last dose (VG161 or nivolumab, calculated at the later of the day).
12. Female patients of childbearing age must have a negative blood pregnancy test within 1 day prior to enrollment.

Exclusion Criteria:

- (Any of the following criteria must be excluded)

1. received chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor drugs within 4 weeks before the first use of the study drug, of which oral fluorouracil and small molecule targeted drugs were within 2 weeks before the first use of the study drug or within 5 half-lives of the drug (whichever was longer).
2. received other unmarketed clinical trial treatment within 4 weeks before the first dose of study drug.
3. Major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks before the first dose of study drug.
4. Patients who have received systemic corticosteroids (prednisone > 10 mg/day or equivalent doses of the same class of drugs) or other immunosuppressive agents within 14 days before the first dose of study drug; except for the following: topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term corticosteroids (≤ 10 mg prednisone equivalent) for prophylaxis (e.g., prevention of contrast agent allergy).
5. Vaccination within 4 weeks prior to the first dose of study drug.
6. Adverse reactions of previous anti-tumor treatment have not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except alopecia and other toxicities judged by the investigator as having no safety risk).
7. Patients with central nervous system metastasis, spinal cord metastasis and/or spinal cord compression.
8. patients with active diverticulitis or symptomatic gastrointestinal ulcers;
9. in the herpes simplex virus recurrence infection period, and there are corresponding clinical manifestations, such as oral herpes labialis, herpes keratitis herpeticum, genital herpes, etc., or there are herpes infection-related complications (herpes keratitis, encephalitis, nerve injury, etc.), and intermittent or long-term use of anti-herpes drugs (e.g., acyclovir) treatment, except intermittent local use.
10. other active uncontrolled infections.
11. History of immunodeficiency, including positive HIV antibody test and positive Treponema pallidum antibody test.
12. Patients with active chronic hepatitis B or active hepatitis C (except hepatitis B virus carriers, stable hepatitis B after drug treatment [HBV-DNA test negative or < 50 IU/ml] and cured hepatitis C patients [HCV RNA test negative]);
13. history of serious cardiovascular disease: 1) ventricular arrhythmia requiring clinical intervention; 2) QTc interval > 480 ms; 3) Acute coronary syndrome, congestive heart failure, stroke or other Grade III or higher cardiovascular events within 6 months; 4) New York Heart Association (NYHA) functional classification ≥ II or left ventricular ejection fraction (LVEF) < 40%; 5) uncontrolled hypertension after treatment (as judged by the investigator).
14. Patients with active, or have had and have had autoimmune diseases that may recur (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes, etc.); but excluding patients with clinically stable autoimmune thyroiditis, autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; type I diabetes using stable doses of insulin; vitiligo or recovered childhood asthma/allergy, and patients who do not require any intervention in adulthood.
15. Having received immunotherapy and have experienced immune-related adverse events (irAEs) such as immune-related pneumonia and myocarditis, which may affect the safety of the investigational drug as judged by the investigator.
16. Patients who have received immune checkpoint inhibitors and develop serious adverse reactions after treatment and need to be permanently disabled.
17. Known alcohol or drug dependence.
18. Mental disorders or poor compliance.
19. Pregnant or lactating women.
20. subjects with pleural effusion or pericardial effusion or ascites requiring clinical intervention.
21. The investigator believes that the subject has other serious systemic diseases or other reasons and is not suitable for this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase Ib:RP2D/MTD | through Phase Ib study completion, an average of 1 year
  RP2D/MTD for VG161 in Combination with Nivolumab
Phase Ib:Incidence and number of DLT | through Phase Ib study completion, an average of 1 year
  Incidence and number of DLT (dose-limiting toxicity)
Phase Ib and Phase IIa:AE, SAE occurrence and frequency | through Phase Ib and Phase IIa study completion, an average of 2 year
  Occurrence and frequency of AE (Adverse Event) and SAE（Serious adverse event)
Phase IIa:ORR | through Phase IIa study completion, an average of 1 year
  Objective response rate (ORR)

SECONDARY OUTCOMES:
Phase Ib and Phase IIa:ORR and DCR | through Phase Ib and Phase IIa study completion, an average of 2 year
  Objective response rate (ORR) and disease control rate (DCR)
Phase Ib and Phase IIa:PFSand OS | through Phase Ib and Phase IIa study completion, an average of 2 year
  Progression Free Survival (PFS) and Overall Survival (OS)
Phase Ib and Phase IIa:DOR | through Phase Ib and Phase IIa study completion, an average of 2 year
  Duration of Response (DOR)
Phase Ib and Phase IIa: Immunological indicators | through Phase Ib and Phase IIa study completion, an average of 2 year
  Immunological parameters: peripheral blood lymphocyte subsets (CD3 +, CD4 +, CD8 +, CD4 +/CD8 + ratio, CD19 +, CD16 + CD56 + (NK) cells), cytokines (IL-12, IL-15, IL-6, TNF-α, IFN-γ);
Phase Ib and Phase IIa:Correlation of PD-L1 combined positive score (CPS) with safety and efficacy | through Phase Ib and Phase IIa study completion, an average of 2 year
  Correlation of PD-L1 combined positive score (CPS) with safety and efficacy
Phase Ib and Phase IIa:Correlation of herpes simplex virus type I antibodies with safety and efficacy | through Phase Ib and Phase IIa study completion, an average of 2 year
  Correlation of herpes simplex virus type I antibodies with safety and efficacy
Phase Ib and Phase IIa:Immunohistochemical detection of HER2、CD68、 CD3、 CD4、 CD8、CD47 | through Phase Ib and Phase IIa study completion, an average of 2 year
  Immunohistochemical detection of HER2、CD68、 CD3、 CD4、 CD8、CD47
Phase Ib :Pharmacokinetic parameters: Blood concentrations of VG161 at different time points after single and multiple doses | through Phase Ib study completion, an average of 1 year
  Pharmacokinetic parameters: Blood concentrations of VG161 at different time points after single and multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No